CLINICAL TRIAL: NCT06957691
Title: Proof-of-Concept Trial to Assess the Efficacy and Safety of Fezolinetant in Improving Vasomotor Symptoms in Men With Prostate Cancer Undergoing Androgen Deprivation Therapy (Fezo-ADT Trial)
Brief Title: Proof-of-Concept Trial to Assess the Efficacy and Safety of Fezolinetant in Improving Vasomotor Symptoms in Men With Prostate Cancer Undergoing Androgen Deprivation Therapy
Acronym: Fezo-ADT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shehzad Basaria, M.D. (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Shehzad Basaria, M.D., Professor of Medicine, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1000264
Record Dates: First submitted 2025-04-14; First posted 2025-05-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Prostate Cancer (Adenocarcinoma); Prostate Cancer Metastatic Disease; Prostate Cancer Recurrent; Prostate Carcinoma; Prostate Neoplasm; Prostate Adenocarcinoma; Prostate Cancer With Bone Metastasis; Vasomotor Disturbance; Vasomotor Symptoms; Vasomotor Symptoms (VMS); Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men; Vasomotor Symptoms; Hot Flashes; Androgen Deprivation Therapy; Androgen Ablative Therapy of Advanced Hormone-dependent Prostate Carcinoma; Androgen-deprivation Therapy; Hot Flashes; Hot Flushes; Hot Flushes and/or Sweats
Keywords: Androgen Deprivation Therapy; Hot Flashes; Hot Flushes; Prostate Cancer; Vasomotor Symptoms
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Multiple Endocrine Neoplasia Type 1; Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fezolinetant (Experimental): Daily oral administration at a dose of 45 mg
  Interventions: Drug: fezolinetant - reference formulation
- Placebo (Placebo Comparator): Daily oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fezolinetant - reference formulation — Daily oral administration of fezolinetant at a dose of 45 mg
  Arms: Fezolinetant
Drug: Placebo — Daily oral administration of placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if fezolinetant can treat hot flashes (vasomotor symptoms) in men with prostate cancer undergoing androgen deprivation therapy.

The main questions it aims to answer are:

* Does fezolinetant improve the frequency and severity of hot flashes?
* Does fezolinetant cause any harm to the liver?
* Does fezolinetant improve quality of life, sleep quality, fatigue, mood, sexual function, and metabolic parameters?

Researchers will compare how people respond to fezolinetant versus a placebo, which does not contain any active medicine.

Participants will:

* Take fezolinetant or a placebo every day for 4 weeks
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of the number of times and intensity that they experience hot flashes

DETAILED DESCRIPTION:
Prostate cancer is the most common type of cancer in men. At the time of initial diagnosis, most men have disease that is confined to the prostate and are typically managed through surveillance or local treatments, such as prostatectomy or radiation therapy. Since the prostate relies on androgens (male hormones), androgen deprivation therapy is the primary treatment for patients with locally advanced, recurrent, or metastatic prostate cancer.

Androgen deprivation therapy involves suppressing the production of androgens in men, which can be achieved through orchiectomy (removal of the testes) or medications like gonadotropin-releasing hormone agonists or antagonists that lower serum testosterone levels to a castrate range (less than 20 ng/dL). In men, 95% of serum estrogen comes from the aromatization of testosterone. Consequently, androgen deprivation not only leads to androgen deficiency but also results in near-absolute estrogen deficiency. The absence of sex hormones in these patients can cause numerous adverse effects, including sexual dysfunction, and loss of muscle and bone. Among these side effects, vasomotor symptoms (such as hot flashes) are particularly debilitating. These symptoms are characterized by sudden feelings of intense heat that spread throughout the body, prompting the activation of heat-dissipation mechanisms to lower body temperature.

Hot flashes are reported by 70-80% of men undergoing androgen deprivation therapy, typically beginning a few weeks after treatment starts, with most men experiencing more than five episodes daily. These vasomotor symptoms significantly affect the patient's quality of life, sleep quality, concentration, and overall productivity. Despite the burden they impose, effective treatments for hot flashes in men undergoing androgen deprivation therapy are still lacking.

The introduction of neurokinin 3 (NK3) receptor antagonists has brought hope to this area. Fezolinetant is a selective NK3 receptor antagonist that has recently been approved for treating moderate to severe vasomotor symptoms in menopausal women. Given that the underlying cause of vasomotor symptoms in both menopausal women and men on androgen deprivation therapy stems from estrogen deficiency, fezolinetant offers an opportunity to assess its efficacy and safety for male patients.

No previous studies have evaluated the effectiveness of NK3 receptor antagonists on vasomotor symptoms in men undergoing androgen deprivation therapy for prostate cancer. Since prostate cancer is the most prevalent solid tumor in men and vasomotor symptoms are common, distressing, and highly burdensome, a trial demonstrating the safety and efficacy of fezolinetant could provide clinicians and patients with a novel, effective, safe, and easy-to-administer treatment that has the potential to transform care for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 40 years and older
* Diagnosis of prostate cancer
* Androgen deprivation therapy
* Presence of 5 or more hot flashes a day that are considered moderate to severe
* Ability to sign the inform consent
* Willing to use reliable methods of contraception if partner is of childbearing age
* Ability to record hot flashes electronically

Exclusion Criteria:

* Use of abiraterone acetate
* Use of docetaxel and other chemotherapeutic agents
* Liver cirrhosis
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) above the upper limit of normal
* Total bilirubin above the upper limit of normal
* Glomerular filtration rate < 30 mL/min
* Use of selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, tricyclic antidepressants, sedatives, or hypnotics
* Use of over-the-counter hormonal agents or herbal compounds
* Current use of CYP1A2 inhibitors
* Ingestion of alcohol within 2 weeks prior to the baseline visit
* Inability to abstain from alcohol use during the study period.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Frequency of Vasomotor Symptoms Through Daily Hot Flash Diary from Baseline to 4 Weeks | From baseline to the end of treatment at 4 weeks.
  Participants achieved a response if they had a significant decrease in scores in the hot flash diary.
Hepatic safety, as assessed by measuring liver function tests | From baseline to the end of treatment at 4 weeks.
  Fezolinetant was considered safe if liver function tests did not change significantly.

SECONDARY OUTCOMES:
Change in quality-of-life symptoms related to hot flashes, as assessed using the Hot Flash-Related Daily Interference Scale | From baseline to the end of treatment at 4 weeks.
  The Hot Flash-Related Daily Interference Scale scores range from 0 to 10, with higher scores meaning a worse outcome. Participants improved if they had a significant decrease in their Hot Flash-Related Daily Interference Scale scores.
Change in overall quality of life, as assessed using the Short Form-36 questionnaire | From baseline to the end of treatment at 4 weeks.
  The Short Form-36 scores range from 0 to 100, with higher scores meaning a better outcome. Participants improved if they had a significant increase in their Short Form-36 scores.
Change in sleep quality, as assessed using the Patient-Reported Outcomes Measurement Information System Sleep Disturbance questionnaire | From baseline to the end of treatment at 4 weeks.
  The Patient-Reported Outcomes Measurement Information System Sleep Disturbance scores range from about 30 to 80, with lower scores meaning better outcome. Patients improved if they had a significant decrease in Patient-Reported Outcomes Measurement Information System Sleep Disturbance scores.
Change in mood, as assessed using the Positive and Negative Affect Schedule questionnaire | From baseline to the end of treatment at 4 weeks.
  The Positive and Negative Affect Schedule questionnaire measures two dimensions of mood, Positive Affect and Negative Affect. The scores in each dimension range from 10 to 50. A higher score in the Positive Affect dimension means a better outcome, and a higher score in the Negative Affect dimension means a worse outcome. Participants improved if they had a significant increase in the Positive Affect dimension scores and a significant decrease in the Negative Affect dimension scores in the Positive and Negative Affect Schedule questionnaire.
Change in sexual function, as assessed using the Sexual Arousal, Interest and Drive questionnaire | From baseline to the end of treatment at 4 weeks.
  The Sexual Arousal, Interest and Drive questionnaire scores range from 0 to 100, with higher scores meaning better outcome. Participants improved if they had a significant increase in Sexual Arousal, Interest and Drive scores.
Change in inflammatory status, as assessed by measuring high-sensitivity C-reactive protein (hsCRP) levels | From baseline to the end of treatment at 4 weeks.
  Participants improved if they had a significant decrease in high-sensitivity C-reactive protein (hsCRP) levels.
Change in fatigue, as assessed using the using the Hypogonadism Energy Diary questionnaire | From baseline to the end of treatment at 4 weeks.
  The Hypogonadism Energy Diary scores range from 0 to 100, with higher scores meaning better outcome. Participants improved if they had a significant increase in Hypogonadism Energy Diary scores.
Change in fatigue, as assessed using the using the Functional Assessment of Chronic Illness Therapy - Fatigue questionnaire | From baseline to the end of treatment at 4 weeks.
  The Functional Assessment of Chronic Illness Therapy - Fatigue scores range from 0 to 160, with higher scores meaning better outcome. Participants improved if they had a significant increase in Functional Assessment of Chronic Illness Therapy - Fatigue scores.
Change in fasting glucose level | From baseline to the end of treatment at 4 weeks.
  Participants improved if they had a significant decrease in fasting glucose level.
Change in glycated hemoglobin (HbA1c) level | From baseline to the end of treatment at 4 weeks.
  Participants improved if they had a significant decrease in glycated hemoglobin (HbA1c) level.
Change in fasting lipid levels | From baseline to the end of treatment at 4 weeks.
  Participants improved if they had a significant decrease in fasting lipid levels.

CONTACTS AND LOCATIONS:
Overall Officials: Shehzad S Basaria, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johnson KA, Martin N, Nappi RE, Neal-Perry G, Shapiro M, Stute P, Thurston RC, Wolfman W, English M, Franklin C, Lee M, Santoro N. Efficacy and Safety of Fezolinetant in Moderate to Severe Vasomotor Symptoms Associated With Menopause: A Phase 3 RCT. J Clin Endocrinol Metab. 2023 Jul 14;108(8):1981-1997. doi: 10.1210/clinem/dgad058. PMID 36734148
- [Background] Lederman S, Ottery FD, Cano A, Santoro N, Shapiro M, Stute P, Thurston RC, English M, Franklin C, Lee M, Neal-Perry G. Fezolinetant for treatment of moderate-to-severe vasomotor symptoms associated with menopause (SKYLIGHT 1): a phase 3 randomised controlled study. Lancet. 2023 Apr 1;401(10382):1091-1102. doi: 10.1016/S0140-6736(23)00085-5. Epub 2023 Mar 13. PMID 36924778
- [Background] Patel B, S Dhillo W. Menopause review: Emerging treatments for menopausal symptoms. Best Pract Res Clin Obstet Gynaecol. 2022 May;81:134-144. doi: 10.1016/j.bpobgyn.2021.10.010. Epub 2021 Nov 17. PMID 34965909
- [Background] Sharma P, Wisniewski A, Braga-Basaria M, Xu X, Yep M, Denmeade S, Dobs AS, DeWeese T, Carducci M, Basaria S. Lack of an effect of high dose isoflavones in men with prostate cancer undergoing androgen deprivation therapy. J Urol. 2009 Nov;182(5):2265-72. doi: 10.1016/j.juro.2009.07.030. Epub 2009 Sep 16. PMID 19758646
- [Background] Harle LK, Maggio M, Shahani S, Braga-Basaria M, Basaria S. Endocrine complications of androgen-deprivation therapy in men with prostate cancer. Clin Adv Hematol Oncol. 2006 Sep;4(9):687-96. PMID 17099626
- [Background] Hunter MS, Stefanopoulou E. Vasomotor symptoms in prostate cancer survivors undergoing androgen deprivation therapy. Climacteric. 2016;19(1):91-7. doi: 10.3109/13697137.2015.1125460. Epub 2015 Dec 16. PMID 26673756
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Lee A. Fezolinetant: First Approval. Drugs. 2023 Aug;83(12):1137-1141. doi: 10.1007/s40265-023-01917-1. PMID 37462862
- [Background] Rance NE, Young WS 3rd. Hypertrophy and increased gene expression of neurons containing neurokinin-B and substance-P messenger ribonucleic acids in the hypothalami of postmenopausal women. Endocrinology. 1991 May;128(5):2239-47. doi: 10.1210/endo-128-5-2239. PMID 1708331
- [Background] Modi M, Dhillo WS. Neurokinin 3 Receptor Antagonism: A Novel Treatment for Menopausal Hot Flushes. Neuroendocrinology. 2019;109(3):242-248. doi: 10.1159/000495889. Epub 2018 Nov 30. PMID 30504731
- [Background] Depypere H, Lademacher C, Siddiqui E, Fraser GL. Fezolinetant in the treatment of vasomotor symptoms associated with menopause. Expert Opin Investig Drugs. 2021 Jul;30(7):681-694. doi: 10.1080/13543784.2021.1893305. Epub 2021 Jul 12. PMID 33724119
- [Background] Skorupskaite K, George JT, Veldhuis JD, Millar RP, Anderson RA. Neurokinin 3 Receptor Antagonism Reveals Roles for Neurokinin B in the Regulation of Gonadotropin Secretion and Hot Flashes in Postmenopausal Women. Neuroendocrinology. 2018;106(2):148-157. doi: 10.1159/000473893. Epub 2017 Apr 5. PMID 28380486
- [Background] Stearns V. Management of hot flashes in breast cancer survivors and men with prostate cancer. Curr Oncol Rep. 2004 Jul;6(4):285-90. doi: 10.1007/s11912-004-0037-y. PMID 15161582
- [Background] Guise TA, Oefelein MG, Eastham JA, Cookson MS, Higano CS, Smith MR. Estrogenic side effects of androgen deprivation therapy. Rev Urol. 2007 Fall;9(4):163-80. PMID 18231613
- [Background] Naoe M, Ogawa Y, Shichijo T, Fuji K, Fukagai T, Yoshida H. Pilot evaluation of selective serotonin reuptake inhibitor antidepressants in hot flash patients under androgen-deprivation therapy for prostate cancer. Prostate Cancer Prostatic Dis. 2006;9(3):275-8. doi: 10.1038/sj.pcan.4500891. Epub 2006 Jun 20. PMID 16786037
- [Background] Russell N, Hoermann R, Cheung AS, Ching M, Zajac JD, Handelsman DJ, Grossmann M. Short-term effects of transdermal estradiol in men undergoing androgen deprivation therapy for prostate cancer: a randomized placebo-controlled trial. Eur J Endocrinol. 2018 May;178(5):565-576. doi: 10.1530/EJE-17-1072. Epub 2018 Mar 16. PMID 29549104
- [Background] Freedland SJ, Eastham J, Shore N. Androgen deprivation therapy and estrogen deficiency induced adverse effects in the treatment of prostate cancer. Prostate Cancer Prostatic Dis. 2009;12(4):333-8. doi: 10.1038/pcan.2009.35. Epub 2009 Sep 1. PMID 19901933
- [Background] Sharifi N, Gulley JL, Dahut WL. Androgen deprivation therapy for prostate cancer. JAMA. 2005 Jul 13;294(2):238-44. doi: 10.1001/jama.294.2.238. PMID 16014598
- See also: Highlights of Prescribing Information. VEOZAH® (fezolinetant) tablets, for oral use. Approval: 2023. Revised: 12/2024 — https://www.astellas.com/us/system/files/veozah_uspi.pdf